CLINICAL TRIAL: NCT01759095
Title: Electronic Multidrug Blister Packs to Improve Clinical and Humanistic Outcomes in Patients After Hospital Discharge
Brief Title: Multidrug Blister Pack Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with patient recruitement
Sponsor: Kurt Hersberger (Other)
Responsible Party: Sponsor-Investigator, Kurt Hersberger, Professor PhD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EKBB54/12
Record Dates: First submitted 2012-11-02; First posted 2013-01-02 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Any Event Leading to Hospitalisation
Keywords: adherence; electronic monitoring; primary care; community pharmacy; multidrug blister pack; pill box

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): At hospital discharge, patients of the control group will receive usual care at their community pharmacy.
- Electronic Multidrug Blister Pack (Experimental)
  Interventions: Device: Electronic multidrug blister pack

INTERVENTIONS:
Device: Electronic multidrug blister pack — At hospital discharge, patients will get their prescribed drugs repackaged in an electronic multidrug blister pack with 7x4 cavities. The electronic film affixed on the rear side measures the date and time when a loop is broken, i.e. when a cavity is emptied. Patients will get feedback on their adherence profiles at the community pharmacy.
  Other Names: Multidrug blister pack: Pharmis GmbH, Beinwil am See, Switzerland; Electronic film: Confrérie Clinique S.A., Lausanne, Switzerland
  Arms: Electronic Multidrug Blister Pack

SUMMARY:
The purpose of this study is to determine the benefit of patients using a multidrug blister packs after discharged from an university hospital to their homes.

DETAILED DESCRIPTION:
Typical adherence rates for oral prescription medications are approximately 50-76%. Insufficient adherence causes an increase in morbidity, mortality, and costs, and decreases quality of life of patients. Multidrug blister packs are recommended to improve adherence and are widely used in Switzerland. However, evidence is poor and patient-relevant endpoints are seldom measured. This study was designed to compare patient-relevant outcomes in patients with medication repackaged in multidrug blister packs versus patients with medication dispensed in commercially available packages. Adherence of the intervention group will be monitored electronically and feedback will be given to the patients. The intervention will take place in a study pharmacy. Follow-up visits will take place at the study pharmacy at 3, 6, and 12 months for all patients. Study duration will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Prescription of 4 or more different oral solid drugs
* Capable to understand german (verbally and written)
* Capable to give informed consent
* Insured by a Swiss health insurance
* Manages his/her pharmacotherapy without external support
* Obtains his/her medication from a community pharmacy
* Accepts to use an electronic multidrug blister pack
* Place of domicile in Basel-Stadt or Basel-Land

Exclusion Criteria:

* Pregnancy
* > 2 drugs that cannot be packed into a multidrug blister pack (e.g. fluids)
* Dementia, or evaluated as cognitively impaired by the responsible nurse
* Transplanted patient
* Anticoagulation with oral vitamin K antagonists
* Has already used a multidrug blister pack of Pharmis or a Medifilm® single dose system
* is visually impaired (blind)
* cannot push drugs through a blister
* refuses to allow contact to his/her regular pharmacy and GP
* is referred to a nursing home or to rehabilitation or another hospital at discharge
* is included in other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to rehospitalisation + time to major therapy adjustment | 12 months
  The outcome measure will be assessed at 3, 6, and 12 months.
Medication Possession Ratio | 12 months
  MPR will be assessed at 3, 6, and 12 months.

SECONDARY OUTCOMES:
Timing and taking adherence according to the electronic monitoring system and through patient self report | 12 months
  Electronic monitoring will be continuous over 12 months. Patient self report will be assessed at 3, 6, and 12 months.
Quality of life | 12 months
  Quality of life will be assessed at 3, 6, and 12 months.
Patient satisfaction | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Prof PhD, Study Chair — University of Basel
Locations (1):
- Notfallapotheke, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Mahtani KR, Heneghan CJ, Glasziou PP, Perera R. Reminder packaging for improving adherence to self-administered long-term medications. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD005025. doi: 10.1002/14651858.CD005025.pub3. PMID 21901694
- [Background] Cramer JA. Enhancing patient compliance in the elderly. Role of packaging aids and monitoring. Drugs Aging. 1998 Jan;12(1):7-15. doi: 10.2165/00002512-199812010-00002. PMID 9467683
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Rosen MI, Rigsby MO, Salahi JT, Ryan CE, Cramer JA. Electronic monitoring and counseling to improve medication adherence. Behav Res Ther. 2004 Apr;42(4):409-22. doi: 10.1016/S0005-7967(03)00149-9. PMID 14998735
- See also: Pharmaceutical Care Research Group, University of Basel, Switzerland — http://www.pharmacare.unibas.ch